CLINICAL TRIAL: NCT02538861
Title: Acute Chest Pain Imaging in Emergency Department With Combined Approach of Coronary CT Angiography and CT Myocardial Perfusion
Brief Title: Acute Chest Pain Imaging in the ED With the Combine CCTA and CT Perfusion
Status: Completed | Type: Observational
Sponsor: Baptist Health South Florida (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB#15-062
Record Dates: First submitted 2015-08-18; First posted 2015-09-02 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain | interventions — Computed Tomography Angiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ARM-A: Arm-A patients will receive the standard of care diagnostic test at Baptist Hospital, which includes SPECT imaging
  Interventions: Diagnostic Test: SPECT Imaging Test at Baptist hospital
- ARM-B (Group-1): Group-1 will receive CT Angiography and CT myocardial perfusion with new Revolution CT scanner.
  Interventions: Diagnostic Test: CT Angiography and CT myocardial perfusion at West Kendall Baptist Hospital
- ARM-B (Group-2): The Group-2 of arm B will receive SPECT imaging test.
  Interventions: Diagnostic Test: SPECT Imaging Test at West Kendall Baptist Hospital

INTERVENTIONS:
Diagnostic Test: SPECT Imaging Test at Baptist hospital — Single Photon Emission Tomography (SPECT) testing at Baptist Hospital.
  Groups: ARM-A
Diagnostic Test: CT Angiography and CT myocardial perfusion at West Kendall Baptist Hospital — The combined approach of CT Angiography and CT myocardial perfusion with new Revolution CT scanner
  Groups: ARM-B (Group-1)
Diagnostic Test: SPECT Imaging Test at West Kendall Baptist Hospital — Single Photon Emission Tomography (SPECT) testing at West Kendall Baptist hospital.
  Groups: ARM-B (Group-2)

SUMMARY:
This is a prospective open label two arms clinical trial. ARM-A patients will receive the standard of care diagnostic test at Baptist Hospital Main (BHM), which includes Single Photon Emission Computed Tomography (SPECT) imaging, while ARM-B patients will be randomized sequentially into two groups; Group-1 will receive CT Angiography and CT myocardial perfusion with new Revolution CT scanner (General Electric Healthcare) while the Group-2 will receive SPECT imaging test; both groups of ARM-B at West Kendall Baptist Hospital (WKBH). The primary hypothesis is that the combined evaluation of CT angiography with CT myocardial perfusion is more efficient in detecting or excluding acute coronary syndrome resulting in early discharge and decrease length of stay of patients from the Emergency Department (ED) compared to a strategy with SPECT alone. The secondary hypothesis is that a strategy with CTA/CTP can reduce direct patient care costs and potentially improve patient outcomes in the same patient population when compared to a strategy with SPECT imaging alone.

The main purpose of this study is to have a definite ED chest pain admission triage, which will help to reduce the length of stay and direct patient cost. This approach will reduce the economic burden in intermediate risk group patients as well. We had a Baptist statistician run the numbers. This study will provide important preliminary data to guide clinical implementation of CTP/CTA in clinical practice. We divided arm B into two groups as the CT protocol might be different at each hospital, so we want to reduce bias as a result of variation in clinical patterns in the different hospitals. Also, we kept 50 patients in arm A (Baptist hospital) to have a control group at the hospital level.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE:

Due to the subjectivity of clinical symptoms and the indirect nature of established ischemia tests, effective initial triage of patients in the ED with acute new onset chest pain is difficult and leads to a high number of patients that are admitted to the hospital despite not having obstructive coronary disease. In the subsequent work up, these patients require extensive testing with significant resource consumption and sometimes delayed treatment. The ability to obtain information on the presence of coronary artery stenoses and plaque early in a noninvasive fashion could substantially enhance initial triage in the ED for these patients.

A combined approach as proposed here using CT coronary angiography to assess the coronary morphology together with CT myocardial perfusion assessment would address morphology and function and help to more correctly characterize coronary lesions for decision making of a potential coronary intervention.

Coronary CTA Analysis:

MDCT data sets are assessed qualitatively for the presence of coronary disease within all coronary segments, including side branches. The assessment is performed on original axial source images; thin slice (5mm) MIP's and MPR reconstructions orthogonal and perpendicular to the vessel centerline, and short axis cross-sectional reconstructions (0.625-mm-thickness). The analysis is performed per segment and per patient.

CT Myocardial Perfusion Analysis:

The initial evaluation of perfusion is performed by reconstruction of short axis images viewed in thick multiplanar reformation (MPR) with slice thickness between 5mm and 10mm. Increasing slice thickness increases the voxel size and thus decrease image noise and improves low contrast resolution. For scans with increased image noise, a smoother reconstruction algorithm is also useful. A true perfusion defect will persist throughout multiple different phases and will be visualized in both systole and diastole. On the other hand, a potential defect that is only present in one phase (i.e. only in systole) and then disappears is likely to represent an artifact due to motion (e.g. false positive). In order to identify regions of myocardium that have minor discrepancies in tissue density, narrow window width is preferred, as higher contrast will be achieved. Measuring the attenuation value on first pass computed tomography (CT) perfusion images is helpful in identifying perfusion defects (HU ~ 50) vs. normal (remote) myocardium (Hounsfield Units (HU) ~ 100). A 17-segment model as defined by the American College of Cardiology (ACC) / American Heart Association (AHA) is used to determine perfusion defect in a particular myocardial segment and coronary artery distribution. A score on a scale from 0-4 is graded for each myocardial segment depending on the extent or area of perfusion defect within the segment. The sum of all the segment scores is used to determine if the patient has a disease (e.g., if the maximum score attainable is 68, so any sum score > 3 correlates to a 5% volume ischemia in the myocardium and is designated as disease at the patient level.)

* Decision to do CT myocardial Perfusion will be made by the cardiac radiologist after the acquisition of the calcium score or after identifying a moderate stenosis or non-evaluable segment as described in the protocol.
* The results of the coronary CT angiography and the CT myocardial Perfusion will be used together to make the decision of whether to send the patient home or to cath. Patients will be admitted for further cardiac investigation if: stenosis > 70% by Coronary CT angiography or intermediate stenosis (50-70%)/non-diagnostic resting coronary CT angiography with CT myocardial perfusion defect. Patients will be considered negative and excluded from acute coronary syndrome if stenosis by coronary CT angiography is < 50% or an intermediate/non-diagnostic lesion is seen and no myocardial ischemia is present by CT myocardial Perfusion.

Study Objective The main purpose of this study is to have a definite ED chest pain admission triage, which will help to reduce the length of stay and direct patient cost. This approach will reduce the economic burden in intermediate risk group patients as well.

Study Hypotheses

The proposed study seeks to evaluate the following hypotheses:

I- The combined evaluation of CT angiography with CT myocardial perfusion is more efficient in correctly diagnosing the obstructive disease. This will reduce the length of hospital stay (LOS), in the assessment of intermediate risk patients at detecting or excluding acute coronary syndrome, in patients presenting with chest pain to ED as compared to a strategy with SPECT alone.

II- To reduce the direct patient care costs in the same patient population. This study is proposing a new chest pain algorithm in arm-B at West Kendall Baptist hospital (combined approach of CT angiography and CT myocardial perfusion) that will reduce the length of stay as well as the consumed resources in comparison with the current approach. The additional value of CT myocardial perfusion is to avoid false positive results by CT angiography alone. CT myocardial perfusion will also provide incremental diagnostic value over and above CT angiography.

STUDY DESIGN

This is a prospective open label two-arm clinical trial. Arm-A patients will receive the standard of care diagnostic test at Baptist Hospital, which includes SPECT imaging, while Arm-B patients will be randomized sequentially into two groups; Group-1 will receive CT Angiography and CT myocardial perfusion with new Revolution CT scanner (General Electric Healthcare) while the Group-2 will receive SPECT imaging test; both groups of ARM-B at West Kendall Baptist Hospital. The study population will include a total of 250 patients presenting at the ED with an episode of new onset chest pain. Both study arms will use the 5-Level Miami Baptist Chest Pain Protocol for triage in the ED. This chest pain protocol will be used as previously published at Baptist Hospital and patients triaged there will serve as a reference population (n=50), while patients (n=100) presenting at the West Kendall Baptist Hospital will be triaged using a modified chest pain protocol which includes coronary CT angiography and CT myocardial perfusion assessment at protocol Level 3 (and selected level 4) instead of SPECT (Group-1) and patients (n=100) at West Kendall Baptist Hospital will receive SPECT imaging test (Group-2). The same group of doctors will provide the interpretation for both arms for SPECT images. All the CT scan data (including SPECT imaging, CT Angiography, and CT myocardial perfusion) are transferred to PACS, which is a system of storing the data electronically and can be accessed by the Radiologist. The Radiologist will be blinded to the research patient data.

The study coordinator will collect the study data including; patient length of stay, direct cost and CT scan data related to chest pain episode. Those patients who are discharged from the ED will be contacted by a telephone call after 30 days for a follow-up of MACE event. In case the patient is not available and there is no source of contact information, their medical records will be checked or their primary care doctor will be contacted.

STUDY PROCEDURES

Patient screening will occur at the time when a patient presents at the ED of either hospital and is assigned a categorizing level based on the 5-Level Miami Baptist Chest Pain Protocol. Patients with an assigned "Level 3 and Level 4", who will meet all the inclusion and none of the exclusion criteria, will be invited to participate in the study.

Informed Consent

Once the Investigator or study coordinator has determined the patient's eligibility for the study, the background of the proposed study, the benefits and risks of the procedures will be explained to the patient. All potential patients must agree and sign informed consent documents prior to performing any study-specific procedures including any pre-medications. Patients enrolled at Baptist Hospital will be treated according to the current standard of care practice. They are being asked to consent simply according to privacy law to allow the use of their data for further scientific evaluation. Patients enrolled at West Kendall Baptist Hospital will consent to be treated according to a modified 5-Level Miami Baptist Chest Pain Protocol, in which a SPECT nuclear perfusion scan is replaced by a coronary CT angiography and a CT myocardial perfusion study for Level 3 patients, and a CT myocardial perfusion study is added for Level 4 patients, with intermediate stenoses (40-70%), Agatston Calcium Score >400, or non-evaluable segments in CT angiography due to calcifications, motion artifacts, or technical reasons. Patient in ARM-B will be randomized sequentially and divided into two groups; group-1 will receive the CT Angiography and CT myocardial perfusion while group-2 will receive the SPECT imaging test. Patients at West Kendall Baptist Hospital will provide consent to share their de-identified data with General Electric Healthcare for scientific evaluation, product development, and potential marketing use. Only the West Kendall Baptist hospital revolution study data will be shared with General Electric Healthcare.

DATA MANAGEMENT AND STATISTICAL ANALYSIS:

All the eligible patients will be assigned a study ID and their personal information will be strictly kept confidential. All the data will be collected and analyzed for research purposes. The General Electric heath care will have only access to the West Kendall Arm Revolution Computed tomography patient de-identified data. For statistical analysis, the investigator will do the interim analysis once the enrollment and follow-up call is complete. A biostatistician will independently analyze the data of this protocol.

SAFETY CONSIDERATIONS:

The experience of undergoing computed tomography is not uncomfortable. Computed tomography scanning results in a measurable radiation exposure. Volume coverage of the whole heart with axial mode results in an effective radiation dose of approximately 1 to 10 mSv, comparable to a standard chest multi-detector computed tomography (MDCT) exam (typically 8 to 10 mSv) or nuclear perfusion stress imaging. MDCT requires the injection of iodinated contrast agent. This, in general, poses a risk of renal dysfunction and contrast allergy. The dose of contrast is lower than in the majority of conventional contrast-enhanced computed tomography studies and adequate measures will be taken to identify patients with known contrast allergy or renal dysfunction and exclude them from participation in the study. Administration of Metoprolol (heart beat lowering medication) might lower blood pressure and cause dizziness as well as bronchospasm and allergic reaction. In this case, a physician will provide adequate treatment. Patients that have known contraindications and allergy to Metoprolol are not enrolled. The most common side effects of Regadenoson are shortness of breath, headache, flushing, chest discomfort or chest pain, dizziness, nausea, abdominal discomfort, a metallic taste in the mouth, and feeling hot. Most common side effects began soon after receiving Regadenoson and went away within 15 minutes except for a headache, which is resolved in most patients within 30 minutes

ELIGIBILITY:
Inclusion Criteria:

1. The patient is > 35 years of age.
2. The patient had an episode of chest pain at rest or during exercise within the previous 24 hours.
3. The patient is classified as "Level 3" in the 5-Level Miami Baptist Chest Pain Protocol (Cury R et al. AJR, 2012; 200: 57-65) (44) or The patient is classified as "Level 4" in the 5-Level Miami Baptist Chest Pain Protocol, and has either a 40-70% stenosis by coronary CT angiography, an Agatston Calcium Score >400, or non-evaluable segments in coronary CT angiography due to calcifications, motion artifacts, or other technical reasons. (Level 4 patients who have already been scan for CTA; will not have to repeat the CTA. Eligible Level 4 patients will only go for CT Myocardial Perfusion scan.
4. Women of childbearing potential have a negative pregnancy urine or serum test.
5. The patient understands the study requirements and procedures and provides written informed consent using a form that has been approved by the Institutional Review Board (IRB) before any study specific test or procedures are performed.
6. The patient is willing to comply with the specified follow-up telephone call.

Exclusion Criteria:

1. The patient is classified as "Level 1", "Level 2", or "Level 5" in the 5-Level Miami Baptist Chest Pain Protocol (Cury R et al. AJR, 2012; 200: 57-65). This includes patients with STEMI (Level-1), NSTEMI or Unstable Angina (Level-2) and non-cardiac chest pain patients (Level-5)
2. Known allergy to iodinated contrast agent or creatinine >1.5mmol/L.
3. Atrial Fibrillation, Flutter or irregular heart rhythm.
4. Known history of severe asthma.
5. Body Mass Index (BMI) >45.
6. Patients in unstable conditions.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * > 35 years of age
  * Patient had an episode of chest pain at rest or during exercise within the past 24 hours
  * Patient is classified as Level 3 Baptist Chest Pain Protocol or the patient is classified as "Level 4" and has either a 40-70% stenosis by coronary CT angiography, an Agatston Calcium Score >400, or non-evaluable segments in coronary CT angiography
  * Women of childbearing potential have a negative pregnancy test
  * Patient understands the study requirements and procedures and provides written informed consent before any study specific test or procedures
  * Patient is willing to comply with the specified follow-up telephone call
  Exclusion Criteria:
  * Patient is classified as Level 1, Level 2, or Level 5 in the Miami Baptist Chest Pain Protocol
  * Known allergy to iodinated contrast agent or creatinine >1.5mmol/L
  * Atrial Fibrillation, Flutter or irregular heart rhythm
  * Known history of severe asthma
  * Body Mass Index >45
  * Patients in unstable conditions
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Length of stay | First 24 to 72 hours
  The average length of stay will be calculated in both study arms. Currently patients have 24 hours of stay at hospital in the chest pain observation unit. We expect and propose that with this new study the length of stay will be reduce to less than 14 hours.

SECONDARY OUTCOMES:
Direct patient costs | First 24 to 72 hours
  Direct patient costs will be measured in both study arms

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo C Cury, MD, Principal Investigator — Baptist Health South Florida
Locations (2):
- United States (2):
  - Baptist Hospital of Miami, Miami, Florida
  - West Kendall Baptist Hospital, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cury RC, Nieman K, Shapiro MD, Butler J, Nomura CH, Ferencik M, Hoffmann U, Abbara S, Jassal DS, Yasuda T, Gold HK, Jang IK, Brady TJ. Comprehensive assessment of myocardial perfusion defects, regional wall motion, and left ventricular function by using 64-section multidetector CT. Radiology. 2008 Aug;248(2):466-75. doi: 10.1148/radiol.2482071478. PMID 18641250
- [Result] Habis M, Capderou A, Ghostine S, Daoud B, Caussin C, Riou JY, Brenot P, Angel CY, Lancelin B, Paul JF. Acute myocardial infarction early viability assessment by 64-slice computed tomography immediately after coronary angiography: comparison with low-dose dobutamine echocardiography. J Am Coll Cardiol. 2007 Mar 20;49(11):1178-85. doi: 10.1016/j.jacc.2006.12.032. Epub 2007 Mar 6. PMID 17367662
- [Result] Lessick J, Dragu R, Mutlak D, Rispler S, Beyar R, Litmanovich D, Engel A, Agmon Y, Kapeliovich M, Hammerman H, Ghersin E. Is functional improvement after myocardial infarction predicted with myocardial enhancement patterns at multidetector CT? Radiology. 2007 Sep;244(3):736-44. doi: 10.1148/radiol.2443061397. Epub 2007 Aug 9. PMID 17690323
- [Result] Mahnken AH, Koos R, Katoh M, Wildberger JE, Spuentrup E, Buecker A, Gunther RW, Kuhl HP. Assessment of myocardial viability in reperfused acute myocardial infarction using 16-slice computed tomography in comparison to magnetic resonance imaging. J Am Coll Cardiol. 2005 Jun 21;45(12):2042-7. doi: 10.1016/j.jacc.2005.03.035. PMID 15963407
- [Result] Nieman K, Cury RC, Ferencik M, Nomura CH, Abbara S, Hoffmann U, Gold HK, Jang IK, Brady TJ. Differentiation of recent and chronic myocardial infarction by cardiac computed tomography. Am J Cardiol. 2006 Aug 1;98(3):303-8. doi: 10.1016/j.amjcard.2006.01.101. Epub 2006 Jun 6. PMID 16860013
- [Result] Nieman K, Shapiro MD, Ferencik M, Nomura CH, Abbara S, Hoffmann U, Gold HK, Jang IK, Brady TJ, Cury RC. Reperfused myocardial infarction: contrast-enhanced 64-Section CT in comparison to MR imaging. Radiology. 2008 Apr;247(1):49-56. doi: 10.1148/radiol.2471070332. PMID 18372464
- [Result] Nikolaou K, Sanz J, Poon M, Wintersperger BJ, Ohnesorge B, Rius T, Fayad ZA, Reiser MF, Becker CR. Assessment of myocardial perfusion and viability from routine contrast-enhanced 16-detector-row computed tomography of the heart: preliminary results. Eur Radiol. 2005 May;15(5):864-71. doi: 10.1007/s00330-005-2672-6. Epub 2005 Mar 18. PMID 15776243
- [Result] Rubinshtein R, Miller TD, Williamson EE, Kirsch J, Gibbons RJ, Primak AN, McCollough CH, Araoz PA. Detection of myocardial infarction by dual-source coronary computed tomography angiography using quantitated myocardial scintigraphy as the reference standard. Heart. 2009 Sep;95(17):1419-22. doi: 10.1136/hrt.2008.158618. Epub 2009 Feb 5. PMID 19196731
- [Result] Gerber BL, Rochitte CE, Melin JA, McVeigh ER, Bluemke DA, Wu KC, Becker LC, Lima JA. Microvascular obstruction and left ventricular remodeling early after acute myocardial infarction. Circulation. 2000 Jun 13;101(23):2734-41. doi: 10.1161/01.cir.101.23.2734. PMID 10851212
- [Result] Cury RC, Feuchtner GM, Batlle JC, Pena CS, Janowitz W, Katzen BT, Ziffer JA. Triage of patients presenting with chest pain to the emergency department: implementation of coronary CT angiography in a large urban health care system. AJR Am J Roentgenol. 2013 Jan;200(1):57-65. doi: 10.2214/AJR.12.8808. PMID 23255742